CLINICAL TRIAL: NCT02294747
Title: Trochanteric Hip Fractures (AO A2) Treated With Sliding Hip Screw With or Without Trochanteric Stabilizing Plate - a Randomized Controlled Trial Using Radiostereometry.
Brief Title: Trochanteric Hip Fractures (AO A2) SHS With or Without Trochanteric Stabilizing Plate - Rct Using RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Frede Frihagen, Consultant, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/475/REK SO B
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Hip Fractures; Trochanteric Fractures; Intertrochanteric Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHS without TSP (Active Comparator): Patients with AO 31 A2 trochanteric fractures operated with sliding hip screw without trochanteric stabilization plate.
  Interventions: Device: Sliding Hip Screw without Trochanteric Stabilization Plate
- SHS with TSP (Active Comparator): Patients with AO 31 A2 trochanteric fractures operated with sliding hip screw with trochanteric stabilization plate.
  Interventions: Device: Sliding Hip Screw with Trochanteric Stabilization Plate

INTERVENTIONS:
Device: Sliding Hip Screw with Trochanteric Stabilization Plate
  Other Names: Lateral Stabilizing Plate, Lateral Support Shield
  Arms: SHS with TSP
Device: Sliding Hip Screw without Trochanteric Stabilization Plate
  Arms: SHS without TSP

SUMMARY:
Trochanteric fractures represent about half of the hip fractures (with femoral neck fractures as the other half). Trochanteric hip fractures are almost always treated surgically with internal fixation of the fracture. However there is a debate ongoing for what is the appropriate implant to use. For stable fracture patterns the evidence seems to be in favor of the sliding hip screw, but for the unstable fractures it is more unclear whether to use a intramedullary nail or sliding hip screw with or without a lateral support plate (TSP). The role of the TSP in clinical use remains unclear and very little has been published about this, but it is believed to be an important contributor of stability to the sliding hip screw construct. We are planning a randomized controlled trial on trochanteric hip fractures to establish a method for implanting the tantalum markers, to observe the fracture healing process and to further investigate the role of the TSP.

DETAILED DESCRIPTION:
Trochanteric fractures represent about half of the hip fractures (with femoral neck fractures as the other half), and are almost always treated surgically with internal fixation of the fracture. However, there is an ongoing debate on what is the appropriate implant to use. For stable fracture patterns the evidence seems to be in favour of the sliding hip screw, whereas for the unstable fractures it is unclear whether an intramedullary nail or a sliding hip screw with or without a lateral support plate should be the implant of choice. A series of studies is now planned at Oslo University Hospital in collaboration with Diakonhjemmet Hospital in hope to further clarify this debate. The use of the lateral/trochanteric support plate (TSP) is widespread in some regions (e.g. Norway, Sweden and parts of Britain), but virtually never used other places. The role of the TSP remains unclear and very little has been published on it's use, even though it is believed to be an important contributor of stability to the sliding hip screw construct.

Trochanteric fractures are mainly caused by a direct trauma, i.e mainly a fall from own height in the elderly. The fractures are most often classified using the Müller AO classification or the Evans/Jensen, but several other classification systems also exist. The ideal classification system should be easily applicable, reliable, and aid in treatment decision making.

The treatment of trochanteric fractures comprise perioperative and operative modalities. The perioperative modalities consist among others of medical optimalization preoperatively, early rehabilitation and prevention of new fractures by treating osteoporosis and preventing new falls. The main scope of the current study will, however, be the operative modalities.

Surgery for trochanteric fractures is performed mainly with fracture reduction on a traction table and internal fixation, using either an intramedullary (IM) nail or a sliding hip screw (SHS), both available in various designs from different manufacturers. The latest Cochrane review did not conclude on which implant is the superior. However, among stable fractures there are less reoperations with the SHS, mainly due to peri-implant femoral fractures after operation with an IM nail that. The more unstable fractures, namely the reverse oblique and subtrochanteric fractures, may obtain better results using an intramedullary nail, probably due to less secondary dislocations with resulting varus deformity, shaft-medialization and shortening. The evidence for this is, however, weak and the role of the TSP remains unclear.

Radiostereometry (RSA) is the most precise and accurate method to measure motion in vivo between different segments in orthopaedic research. To do so, radio-opaque tantalum markers are implanted into the bone defining different segments. Stereoradiographs are performed over time to detect movement and monitor the healing (or non healing) process. This movement can be calculated both as translations and rotations. They are ideal to describe and compare the stability of fracture systems. RSA has been used successfully in earlier studies on fracture healing. Due to the high accuracy and precision, RSA yield reliable results with relatively small study-groups. We plan to use RSA to measure fracture dislocation and time to healing in our studies.

The study will be on the function of the trochanteric support plate and it´s ability to prevent secondary dislocation in AO 31 A2 fractures. We will utilize RSA for measurements during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* AO 31-A2
* able to walk independently, aids such as crutches or walker allowed
* able to consent
* fit for surgery with SHS with or without TSP

Exclusion Criteria:

* not willing or able to attain follow up
* previous fracture or surgery with retained metal work in the same hip
* concomitant disease that will shorten life expectancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Fracture displacement during healing measured with radiostereometry | 52 weeks
  Will be measured by RSA postoperatively, before discharge and after 4, 8, 12, 24 and 52 weeks. Total displacement from first reading to the reading showing maximum displacement is the main outcome.

SECONDARY OUTCOMES:
Perioperative blood loss | 1 week
Time of surgery | 1 week
Eq5d | 52 weeks
  Health Related Quality of Life (Hrqol).
Eq5d | 26 weeks
  Hrqol.
Eq5d | 12 weeks
  Hrqol.
Eq5d | 8 weeks
  Hrqol.
Eq5d | 4 weeks
  Hrqol.
Time to union as measured by RSA (cessation of motion) and radiographs | Will be examined at 4, 8, 12, 26 and 52 weeks
  When RSA shows that no motion has happened between two time points the fracture will be regarded as healed at the former time point.
Time to union as measured by plain radiographs and clinical findings | Will be examined at 4, 8, 12, 26 and 52 weeks
  Composite endpoint: Healing defined by obliteration of fracture line radiographically and pain free weight bearing (except lateral pain from hardware), when this occurs the fracture will be considered healed.
Harris Hip Score | 52 weeks
  Will be examined at 4, 8, 12, 26 and 52 weeks
Harris Hip Score | 26 weeks
  Will be examined at 4, 8, 12, 26 and 52 weeks
Harris Hip Score | 12 weeks
  Will be examined at 4, 8, 12, 26 and 52 weeks
Harris Hip Score | 8 weeks
  Will be examined at 4, 8, 12, 26 and 52 weeks
Harris Hip Score | 4 weeks
  Will be examined at 4, 8, 12, 26 and 52 weeks
Postoperative pain (NRS) while in hospital | 1 week
  Pain at mobilization (NRS) at discharge
Timed Up and Go (Tug) test | 4 weeks
Timed Up and Go (Tug) test | 8 weeks
Timed Up and Go (Tug) test | 12 weeks
Timed Up and Go (Tug) test | 26 weeks
Timed Up and Go (Tug) test | 52 weeks
Pain (NRS) | 4 weeks
  Maximum hip pain during the last week
Pain (NRS) | 8 weeks
  Maximum hip pain during the last week
Pain (NRS) | 12 weeks
  Maximum hip pain during the last week
Pain (NRS) | 26 weeks
  Maximum hip pain during the last week
Pain (NRS) | 52 weeks
  Maximum hip pain during the last week
Satisfaction with operated hip (NRS) | 4 weeks
Satisfaction with operated hip (NRS) | 8 weeks
Satisfaction with operated hip (NRS) | 12 weeks
Satisfaction with operated hip (NRS) | 26 weeks
Satisfaction with operated hip (NRS) | 52 weeks
Motion during healing as measured by radiostereometry. | 52 weeks
  Will be measured by RSA postoperatively, before discharge and after 4, 8, 12, 24 and 52 weeks. Pattern and time of secondary displacement will be compared between the treatment groups during the first year postoperatively.
Motion during healing as measured by plain radiographs., | 52 weeks
  The rate and degree of secondary displacement during the first year will be compared between the groups.

OTHER OUTCOMES:
Reoperation for healing problems | 52 weeks
  Any additional surgery addressing healing problems or hardware failure
Mortality | 52 weeks
  Any reason

CONTACTS AND LOCATIONS:
Overall Officials: Frede Frihagen, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Orthopedic Center, Ulleval University Hospital, Oslo
  - Diakonhjemmet Hospital, Oslo